CLINICAL TRIAL: NCT04203953
Title: Impact of a Quality Improvement Intervention to Promote Early Mobilization in Patients in the Trauma ICU
Brief Title: Quality Improvement Intervention to Promote Early Mobilization in Trauma ICU
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201910048RINB
Record Dates: First submitted 2019-12-12; First posted 2019-12-18 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Patients Admitted to the ICU More Than 3 Days Post-onset

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Early mobilization program — Early mobilization will be defined as any active exercise where the patients could assist with the activity using their own muscle strength and control that occurred within the first 7 days of trauma ICU admission and will be intended to maintain or restore overall function as well as being scored using the ICU mobility scale.15 The ICU mobility scale includes rolling, bridging, sitting, standing and walking, and upper and lower limb flexion and extension. In-bed therapies will include active or active-assist range of motion, bridge exercise, quadriceps setting, straight leg raising, rolling exercises and facilitation.

SUMMARY:
Background: Despite the fact that many lines of evidence point to the safety and feasibility of early mobilization in medical or surgical ICUs, there remains limited evidence regarding the efficacy or outcome of mobilizing patients in trauma ICU. Given the lack of published literature or routine protocol for mobilizing this population in our institution, the investigators developed a formal protocol and quality improvement project.

Objective: To determine the flexibility and effects of an early mobilization project in a trauma ICU.

Design: Observational, pre-post design.

Setting: A eight-bed trauma ICU in a medical center in Taipei.

Patients: Critically ill adults admitted to the trauma ICU.

Intervention: This project will involve a routine care baseline phase to promote early mobilization of critically ill patients. The bedside physical therapist (PT) will assess the appropriateness of the activity level throughout the day. The PT will provide guidelines for appropriate activities, with the option to perform more advanced activities using equipment. Early mobilization will be provided once daily 5 days/week during the 30-minute family visiting time.

Outcome: The primary outcome measures will be as follows: (1) the proportion of patients with occupational therapist (OT) and/or PT consultations per ICU days 3, 7 and 14; (2) the time and types of mobilization activities performed at the day of ICU admission, the day of ICU discharge and the day of hospital discharge, including passive and active activities; (3) the Perme intensive care unit mobility score at the day of ICU admission, the day of ICU discharge and the day of hospital discharge; Secondary outcome measures will include the following: (1) the number of times and reasons for suspended activities; (2) mobilization-related adverse events.

Statistical Analysis: Unadjusted comparisons before and after implementation of the project will be performed using chi-square analysis, Fisher exact test, or the Wilcoxon signed rank test, as appropriate. A two-sided p-value less than 0.05 will be used to determine statistical significance.

DETAILED DESCRIPTION:
Background:

Early mobilization is a component of the ABCDE bundle (Awaken from sedation; Breathe independently from ventilator; Choice of sedation; Delirium management; Early mobilization), an interdisciplinary, patient-centered strategy to facilitate evidence-based practices in intensive care unit (ICU) settings. In patients who underwent early mobilization, specific benefits were fewer ventilator days, fewer ICU and hospital days, fewer hospital complications, less sedation and delirium days, and improved in-hospital functional outcomes. Despite the fact that several lines of evidence demonstrated the safety and efficacy of early mobilization in the ICU, studies conducted in neurological or trauma ICU settings are scarce, possibly because of safety considerations such as physiologic instability (hemodynamic or intracranial pressure) and invasive device integrity. It has only recently been suggested that such programs are effective, safe, and potentially beneficial in critically ill neurological patients. Nevertheless, there is no set protocol in place for moving these patients, nor any suggested parameters to monitor.

Evidence regarding early mobilization has been based on reports from general medical and surgical ICU environments, rather than from neurosurgical ICU (NSICU) or trauma ICU settings. In NSICU patients with acute brain injury mostly, safety during mobilization could be compromised because of hemiparesis or hemiplegia, cognitive impairment, tenuous intracerebral pressure and cerebral perfusion, or dislodgement of cerebral monitoring or other indwelling devices. In trauma ICU, trauma patients often have extensive orthopedic and neurosurgical injuries, creating additional barriers to mobility. Little is known about the potential effects of mobilizing patients with acute brain or server injuries admitted to the trauma ICU. In one pre- and post-intervention research study of early mobilization in patients with neurologic injury treated in a ICU, mobility levels increased post-intervention, without adverse events. The results also supported the notion that progressive early mobilization program leads to shorter ICU and hospital length of stay (LOS), fewer patient restraint days, and fewer hospital-acquired infections. Another relevant study showed that implementation of a progressive mobility algorithm was safe and was associated with a higher likelihood of mobilization in the first week after spontaneous intracerebral hemorrhage (ICH) in the neurological ICU. For trauma patients, previous studies demonstrated the safety of a mobility protocol in a trauma and burn ICU and, additionally, showed a decrease in airway, pulmonary, and vascular complications. Results from another study revealed favorable functional outcomes for patients involved in a structured mobility program with physical therapy in the neuro/trauma ICU. Overall, the lack of available evidence highlights the fact that there remains much research to be done regarding early rehabilitation for patients in the trauma ICU and there are specific questions to be answered regarding the timing of intervention, the intensity and the type of exercises.

Previously, in the trauma ICU of National Taiwan University Hospital (NTUH), the referral of patients for physical therapy and mobilization occurred at the discretion of the medical providers with very low the proportion of patients with physical therapist (PT) consultations. Therefore, the overall objective of this quality improvement (QI) project will be to evaluate a structured and interdisciplinary early rehabilitation and progressive mobility protocol for critically ill patients in a trauma ICU.

Purpose： The goals of the project will be to provide a standardized, evidence-based, interdisciplinary mechanism to increase each patient's activity level safely while simultaneously initiating and promoting a culture of mobility. The investigators will also conduct this project to evaluate the effects of this early mobilization program on the outcomes of patients in the trauma ICU.

Intervention： Overview of Project Setting, Design, and Patients The project initiative will be developed using an established and structured QI framework (described below in "QI Process") and evaluate using an observational, pre-post design. A nonprobability, convenience sampling strategy will be used for program evaluation. The setting will be the trauma ICU in National Taiwan University Hospital, 8-bed trauma ICU unit. PT and Occupational therapist (OT) consultations and treatments will be available when ordered by medical providers. Both the assessment method and training program (progressive mobility protocol for all critically ill patients) are current procedure of the early rehabilitation team. The project will be implemented using equipment resources, the Sara Combilizer or Sara Plus (Arjo Huntleigh, GETINGE group).

This study will consist of a retrospective, pre- QI Process period (January 1, 2018, through June 30, 2019) followed by a prospective QI-Process phase (December 31, 2019-December 31, 2022). We conducted a retrospective review covering the period from January 1, 2018, through June 30, 2019, of patients >20 years of age admitted to the trauma ICU (more than 3 days), who were alive more than 7 days after ICU admission. Charts from the first consecutive 100 patients who meet aforementioned criteria will be reviewed retrospectively before implementation of the QI Process by using the daily medical records and daily assessment reports of nursing built into the electronic medical records of NTUH. The prospective population will consist of patients above 20 years old who required trauma ICU admission for three or more days with PT or/with OT consultations from December, 2019, through December 31, 2022.

QI Process The structured QI model of the project initiative will create a change in practice using the "four Es" approach: engage, educate, execute, and evaluate. To achieve this, a collaborative interdisciplinary QI team, the EM Working Group, will be created. Participation in the EM Working Group will be open to all interested the ICU staff. Active participants will include at least one champion from each of the following groups: physicians, nurse practitioners, nurses, OT, PT and rehabilitation physicians. This core group of individuals will meet on a weekly basis over 2 months to plan (engage and educate) the QI project prior to its execution and evaluation. First, champions from the rehabilitation team will conduct focus groups with all stakeholders from their respective disciplines to present the problem and identify trauma ICU -based facilitators and barriers to early mobilization. Explain why the interventions are important. Bedside staff will better understand the importance of mobility if there is a clear understanding that mobility will increase safety, decrease secondary complications and improve outcomes, ultimately shortening hospital stays and cost of care. Second, the rehabilitation team will develop guidelines for mobilization in the trauma ICU based on the feedback provided from the focus groups and prior literature regarding early mobilization. Third, educational resources will be developed for all trauma ICU staff. Finally, the interdisciplinary team will determine valid and feasible outcome measures based on previously published early mobilization QI studies to evaluate performance.

Staff Educational Resources To ensure competence in treating this patient population, literature will be reviewed on the efficacy and safety of early mobilization and interventions. Then, educational resources will be presented in meetings, presentations, or online communications. A formal written procedure will also be available to staff. A relevant online learning module regarding early rehabilitation in critically ill patients will be created.

The Early Mobilization Program Early mobilization will be defined as any active exercise where the patients could assist with the activity using their own muscle strength and control that occurred within the first 7 days of trauma ICU admission and will be intended to maintain or restore overall function as well as being scored using the ICU mobility scale. The ICU mobility scale includes rolling, bridging, sitting, standing and walking, and upper and lower limb flexion and extension. In-bed therapies will include active or active-assist range of motion, bridge exercise, quadriceps setting, straight leg raising, rolling exercises and facilitation. Safety criteria for early mobilization will be evaluated the following before intervention: Glasgow Coma Scale (GCS) above 6; raised intracranial pressure<20mmHg; no cardiopulmonary arrest; no acute myocardial infarction; no rapidly developing neuromuscular disease; no pregnancy; no ruptured or leaking aortic aneurysm; and no ICU admission for palliative care or no medical orders specifying alternate activities.

It does not preclude the patient receiving assistance from staff or equipment. The protocol will include an initial assessment by the physician on service to determine readiness to participate in PT. If deemed appropriate, PT and OT consults will be requested. It will be determined whether each patient's activity level will evaluated by the rehabilitation team. PTs will facilitate active mobility, while range of motion, seating, and positioning will be the purview of PTs, with OT collaboration as needed. The bedside PT will record this information in the electronic record daily performances and goals note. The bedside PT will also assess the appropriateness of the activity level throughout the day by the ICU mobility scale. Activities may be implemented by nurses and/or therapists based on their specific skills and provided equipment. The PT will provide guidelines for appropriate activities, with the option to perform more advanced activities using equipment (Sara Combilizer or Sara Plus) Note: individualized to the patient. PTs will teach the family how to do passive or active range of motion, bed exercises, and sitting position in bed for the patient as well as encourage the family to assist with these exercises when they visit. Early mobilization will be provided once daily 5 days/week during the 30-minute family visiting time (morning or afternoon visits).

Severe adverse events will be prospectively defined as falls, unplanned extubation, cardiac arrest, loss of an invasively-inserted line and new-onset atrial or ventricular tachyarrhythmia; all these will be recorded during mobilization sessions. The investigators will define adverse events that will require a mobilization session to be suspended prematurely a priori. These events include decrease in mean arterial pressure <60 mmHg or decrease in oxygen saturation <88% for more than 3 minutes or occurrence of a new oxygen requirement with a fraction of inspired oxygen >0.6. If an adverse event occurs during a therapy session, the session will be immediately stopped and the attending physician will be notified.

ELIGIBILITY:
Inclusion Criteria:

* patients >20 years of age admitted to the trauma ICU (more than 3 days)
* who were alive more than 7 days after ICU admission

Exclusion Criteria:

* patients < 20 years old who required trauma ICU admission for less than three days
* died after ICU admission
* Glasgow Coma Scale (GCS) < 6
* raised intracranial pressure>20mmHg
* with cardiopulmonary arrest
* with acute myocardial infarction
* with rapidly developing neuromuscular disease
* with pregnancy
* with ruptured or leaking aortic aneurysm
* ICU admission for palliative care or medical orders specifying alternate activities.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with OT and/or PT consultations by ICU | up to 1 year
  on days 3, 7 and 14 after onset
the time mobilization activities performed in the ICU | up to 1 year
  on the day of ICU admission, the day of ICU discharge and the day of hospital discharge
the types of mobilization activities performed in the ICU | up to 1 year
  on the day of ICU admission, the day of ICU discharge and the day of hospital discharge. The activities including passive and active activities.
the Perme intensive care unit mobility score | up to 1 year
  on the day of ICU admission, the day of ICU discharge and the day of hospital discharge. The Perme ICU Mobility Score ranges from 0 to 32. The score is derived from 15 items grouped in 7 categories: mental status, potential mobility barriers, functional strength, bed mobility, transfers, gait, and endurance. The score uses a maximum range of 2 to 4 points for each of the 15 items, and it provides a total score that reflects the patient's mobility status at one particular moment in time. A high score indicates few potential mobility barriers and decreased assistance whereas a low score indicates more potential barriers to mobility and more assistance needed for mobility.

SECONDARY OUTCOMES:
the number of times that activities were stopped | up to 1 year
the reasons that activities were stopped | up to 1 year
mobilization-related adverse events | up to 1 year
  including inadvertent extubation or line removal

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan